CLINICAL TRIAL: NCT05677360
Title: HPV Multilevel Intervention Strategies Targeting Immunization in Community Settings (HPV MISTICS)
Acronym: HPV MISTICS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack or Limited Slot Availability
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Department of Health (Other Government); Health Choice Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: MCC-21902
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Human Papilloma Virus (HPV) Vaccine
Keywords: Human Papillomavirus; Vaccination; Multi-level intervention; Community Health Centers; Behavioral
MeSH Terms: conditions — Papillomavirus Infections; Behavior

STUDY DESIGN:
Intervention Model Description: Hybrid Type 1 implementation design which will allow the team to examine both effectiveness of HPV MISTICS and implementation outcomes in a single study. Implementation outcomes will be evaluated using the RE-AIM Qualitative Evaluation for Systematic Translation (RE-AIM QuEST) framework, a mixed-methods framework to identify implementation barriers and facilitators while assessing implementation outcomes (e.g., reach, adoption, implementation, maintenance/sustainability) with a focus on evaluating equity across these outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wave 1: Initial Community Health Centers (Experimental): Initial group of community health centers to receive intervention
  Interventions: Behavioral: HPV MISTICS -Provider Level; Behavioral: HPV MISTICS - Parent Level; Behavioral: HPV MISTICS- HPV Vaccine Champion Level
- Wave 2: Second Community Health Centers (Experimental): Second group of community health centers to receive intervention
  Interventions: Behavioral: HPV MISTICS -Provider Level; Behavioral: HPV MISTICS - Parent Level; Behavioral: HPV MISTICS- HPV Vaccine Champion Level

INTERVENTIONS:
Behavioral: HPV MISTICS -Provider Level — The HPV MISTICS (Multilevel Intervention Strategies Targeting Immunization in Community Settings) provider-level intervention for all clinical staff (e.g., physicians, nurses, medical assistants) includes a 1-hour online training session on the Announcement Approach (i.e., presumptive recommendation) to recommend adolescent vaccinations.
Behavioral: HPV MISTICS - Parent Level — The HPV MISTICS (Multilevel Intervention Strategies Targeting Immunization in Community Settings) parent-level intervention includes a low literacy pre-visit HPV vaccine notification post card in the parent's preferred language.
Behavioral: HPV MISTICS- HPV Vaccine Champion Level — The HPV MISTICS (Multilevel Intervention Strategies Targeting Immunization in Community Settings) system-level intervention involves training an HPV Vaccine Champion at each FQHC on the provider and parent EBIs to monitor and share clinic HPV initiation and completion rates with providers, and to implement reminder/recall systems for subsequent vaccine doses

SUMMARY:
This intervention study will use parent-, provider-, and health center-level strategies to promote HPV vaccination among 11-17 year olds receiving care in 8 community health centers in Florida, will explore factors related to the intervention effect, and will explore implementation outcomes of the intervention.

DETAILED DESCRIPTION:
The goals of this multi-level intervention study are to: 1) test whether HPV MISTICS intervention increases human papillomavirus (HPV) vaccine initiation and completion rates among 11-17-year-old adolescents in 8 Health Choice Network-affiliated community health centers in Florida. 2) Explore other factors related to the intervention effect. 3) Explore implementation outcomes (i.e., reach, adoption, implementation, maintenance, and sustainability) and identify implementation barriers and facilitators with a focus on equity. The study will use parent-, provider-, and health center-level strategies to promote HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* For Staff:
* 18 years of age or older
* Working within the participating Federally Qualified Health Center system
* Able to read, write and speak English
* For Providers:
* 18 years of age or older
* Working within the participating Federally Qualified Health Center system
* Interacting with parents of adolescents ages 11-17
* Able to read, write and speak English
* For parents:
* Parent of 11-17 year old child that has received care within the prior two months at one of the participating Federally Qualified Health Centers
* Whose child has not initiated or completed the HPV vaccine series at the time of their last visit
* Able to read, write and speak English or Spanish, or Haitian Creole

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: HPV Vaccine series initiation rates | at 5 years
  HPV vaccine series initiation (1st dose) rates among adolescents ages 11-17 will be determined on a monthly basis as well as annually. Providers' vaccination rate data for their patient panel (using Florida SHOTS - a free, statewide centralized online immunization information system) will be compared to the National Immunization Survey-Teen (NIS-TEEN) data for the state of Florida.
Effectiveness: HPV Vaccine series completion rates | at 5 years
  HPV vaccine series completion (2nd and 3rd dose) rates among adolescents ages 11-17 will be determined on a monthly basis as well as annually. Providers' vaccination rate data for their patient panel (using Florida SHOTS - a free, statewide centralized online immunization information system) will be compared to the National Immunization Survey-Teen (NIS-TEEN) data for the state of Florida.

SECONDARY OUTCOMES:
Implementation outcome: Reach | at 5 years
  The intervention's implementation will be evaluated for reach - proportion of eligible patients that receive the intervention.
Implementation outcome: Reach demographics | at 5 years
  The intervention's implementation will be evaluated for reach - demographics of patients reached.
Proportion of Healthcare providers who participate in the intervention | at 5 years
  The proportion of health care providers who participate in the intervention, measured by contact log data.
Proportion of Healthcare Providers, Rural vs Urban | at 5 years
  The proportion of health care providers in rural vs urban Federally Qualified Health Centers in network that participate.
Proportion of Health Care providers who complete training | at 5 years
  The proportion of participating health care providers and staff who complete training per site will be measured using the training attendance log
Intervention Sustainability: Health care Providers | at 5 years
  Long term intervention effects and use over time will be determined semi-structured interviews of providers
Intervention Sustainability: Healthcare staff | at 5 years
  Long term intervention effects and use over time will be determined semi-structured interviews of health care staff.

CONTACTS AND LOCATIONS:
Overall Officials: Susan T Vadaparampil, PhD, MPH, Principal Investigator — Moffitt Cancer Center; Shannon Christy, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- [Derived] Christy SM, Patel L, Arevalo M, Fuzzell L, Whitmer A, Turner K, Gore LR, Chung-Bridges K, Parras D, Endemano EY, Brownstein NC, Vadaparampil ST. HPV Multilevel Intervention Strategies Targeting Immunization in Community Settings (HPV MISTICS): Study protocol for a hybrid 1 stepped-wedge cluster randomized trial. Contemp Clin Trials. 2024 Jul;142:107576. doi: 10.1016/j.cct.2024.107576. Epub 2024 May 17. PMID 38763306